CLINICAL TRIAL: NCT03546764
Title: The Small (14F) Percutaneous Catheter vs. Large (28-40F) Open Chest Tube for Traumatic Hemothorax (P-CAT): A Multi-center Randomized Clinical Trial
Brief Title: Multi-center:The Small (14F) Percutaneous Catheter vs. Large (28-40F) Open Chest Tube for Traumatic Hemothorax (P-CAT)
Acronym: P-CAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1506936985A001
Record Dates: First submitted 2018-03-13; First posted 2018-06-06 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: The Efficacy of Percutaneous Catheter vs. Open Chest Tube; Traumatic Hemothorax
Keywords: Percutatneous catheter; chest tube; trauma; hemothorax
MeSH Terms: conditions — Wounds and Injuries; Hemothorax | interventions — Catheter Ablation; Middle Ear Ventilation

STUDY DESIGN:
Intervention Model Description: Two arms - Percutaneous catheter arm vs Chest tube arm
Who Masked: Participant
Masking Description: Patient does not know the details of the treatment assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Percutaneous Catheter (Experimental): 14-French Percutaneous catheter (pigtail or non-pigtail) placed at bedside using Seldinger technique
  Interventions: Device: Percutaneous catheter
- Chest tube (Active Comparator): Placement of 28-36F chest tube placed at bedside by an open cut-down technique (traditional)
  Interventions: Device: Percutaneous catheter

INTERVENTIONS:
Device: Percutaneous catheter — tube inserted to drain hemothorax
  Other Names: tube insertion

SUMMARY:
After sustaining severe trauma to the chest, patients will often bleed into the chest cavity (pleural space) which is called hemothorax or they may also experience air leakage within the chest cavity in combination with the bleeding (hemopneumothorax). These conditions are treated with the insertion of a tube into the chest called a chest tube (CT). Insertion of the CT is very painful for the patient due to the size or diameter of the tube. Alternative to CT is a small percutaneous catheter (PC), pigtail or non-pigtail. At Banner-University of Arizona Tucson Campus (B-UATC) investigator prefers inserting a small pigtail catheter for the management of hemothorax or hemopnuemothorax. The primary purpose of our study is to see if the use of the PC is just as effective as CT in terms of removing leaked blood and/or air from the chest cavity.

DETAILED DESCRIPTION:
The standard treatment for traumatic hemothorax (HTX) and hemopneumothorax (HPTX) has been an insertion of a large-bore chest tube (CT) (French 28-40). The procedure is associated with significant patient's pain and discomfort. Our institution has taken a lead role to replace chest tube insertion with percutaneous (pigtail) catheter (PC) (14F) insertion. The investigators have previously published that, not only PC works just as well as the traditional CT for both pneumothorax (1) and hemothorax( 2), but it is also associated with a significant less insertion pain and tube site pain (3). In that hemothorax study, investigator reported 36 patients who received PC for HTX (2) with the same success as 32F chest tube in term of initial output and success rate; success rate was defined as no further intervention was needed. Since the completion of that study (December 2011), our division has inserted probably 100 PC for hemothorax and hemopneumohthorax Therefore, investigator now believes that it is time for us to demonstrate the efficacy of the PC for hemothorax with a prospective and randomized study as investigators have done previously for traumatic pneumothorax (3).

The investigator hypothesizes that PC will be just as effective as CT in patients with traumatic HTX and HPTX.

Our study aim is to demonstrate the efficacy of the PC in a prospective and randomized fashion as we have done previously in pneumothorax.

Our primary end point is the success/failure rate. Failure is defined as patient require a second intervention i.e., second tube, video-assisted thoracoscopy (VATS), etc.

Our secondary end points are the amount of initial tube drainage (1-hour), 24-hour, 48-hour, 72-hour; tube insertion-related complications, hospital length of stay, and patient's experience during CT/PC insertion (if patient can provide the information).

Significance of the study:

Currently, most trauma surgeons prefer CT over PC for the management of traumatic HTX. The study will provide a level 1 scientific evidence that PC works as well as CT for traumatic HTX/HPTX, and we have already shown that PC is less painful than CT.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18
2. Traumatic HTX/HPTX requiring chest tube insertion

Exclusion Criteria:

1. Emergent indication, hemodynamic instability
2. Patient refuses to participate
3. Prisoner
4. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Failure rate | 30 days
  Failure rate is defined as any second intervention to treat retained hemothorax

SECONDARY OUTCOMES:
Insertion-related complication | 30 days
  any insertion-related complication, minor or major
Hospital course outcome | 30 days
  ICU length of stay, hospital length of stay

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Ariznoa Medican Center, Main campus, Tucson, Arizona
  - Emory University, Atlanta, Georgia
  - University of Nebrask, Omaha, Nebraska
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bauman ZM, Kulvatunyou N. 14-French Pigtail Catheters for Traumatic Hemothorax/Hemopneumothorax: Size Does Not Matter: Reply. World J Surg. 2018 Aug;42(8):2687-2688. doi: 10.1007/s00268-018-4508-y. No abstract available. PMID 29423739
- [Result] Bauman ZM, Kulvatunyou N, Joseph B, Jain A, Friese RS, Gries L, O'Keeffe T, Tang AL, Vercruysse G, Rhee P. A Prospective Study of 7-Year Experience Using Percutaneous 14-French Pigtail Catheters for Traumatic Hemothorax/Hemopneumothorax at a Level-1 Trauma Center: Size Still Does Not Matter. World J Surg. 2018 Jan;42(1):107-113. doi: 10.1007/s00268-017-4168-3. PMID 28795207
- [Result] Kulvatunyou N, Erickson L, Vijayasekaran A, Gries L, Joseph B, Friese RF, O'Keeffe T, Tang AL, Wynne JL, Rhee P. Randomized clinical trial of pigtail catheter versus chest tube in injured patients with uncomplicated traumatic pneumothorax. Br J Surg. 2014 Jan;101(2):17-22. doi: 10.1002/bjs.9377. PMID 24375295
- [Result] Kulvatunyou N, Joseph B, Friese RS, Green D, Gries L, O'Keeffe T, Tang AL, Wynne JL, Rhee P. 14 French pigtail catheters placed by surgeons to drain blood on trauma patients: is 14-Fr too small? J Trauma Acute Care Surg. 2012 Dec;73(6):1423-7. doi: 10.1097/TA.0b013e318271c1c7. PMID 23188235
- [Result] Kulvatunyou N, Vijayasekaran A, Hansen A, Wynne JL, O'Keeffe T, Friese RS, Joseph B, Tang A, Rhee P. Two-year experience of using pigtail catheters to treat traumatic pneumothorax: a changing trend. J Trauma. 2011 Nov;71(5):1104-7; discussion 1107. doi: 10.1097/TA.0b013e31822dd130. PMID 22071915
- [Derived] Hylands M, Gomez D, Beckett A. Letter to the editor: The small (14 Fr) percutaneous catheter (P-CAT) versus large (28-32 Fr) open chest tube for traumatic hemothorax: A multicenter randomized clinical trial. J Trauma Acute Care Surg. 2022 Sep 1;93(3):e125. doi: 10.1097/TA.0000000000003647. Epub 2022 May 25. No abstract available. PMID 35610739
- [Derived] Kulvatunyou N, Bauman ZM, Zein Edine SB, de Moya M, Krause C, Mukherjee K, Gries L, Tang AL, Joseph B, Rhee P. The small (14 Fr) percutaneous catheter (P-CAT) versus large (28-32 Fr) open chest tube for traumatic hemothorax: A multicenter randomized clinical trial. J Trauma Acute Care Surg. 2021 Nov 1;91(5):809-813. doi: 10.1097/TA.0000000000003180. PMID 33843831